CLINICAL TRIAL: NCT05448716
Title: Longitudinal Changes in Left Atrial Strain and Supraventricular Arrhythmia Burden in Cardiac Light Chain Amyloidosis Patients Following Chemotherapy
Brief Title: Left Atrial Strain and Supraventricular Arrhythmia Burden in Cardiac Light Chain Amyloidosis Following Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Deniz Mutlu, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: 2021-53810
Record Dates: First submitted 2022-07-02; First posted 2022-07-07 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Supraventricular Arrhythmia; Left Atrial Abnormality; Amyloid Cardiomyopathy; Congestive Heart Failure
Keywords: Left atrial strain; Supraventricular Arrhythmia; Heart failure; cardiac amyloidosis; Amyloid Cardiomyopathy; Arrhythmia; Strain Imaging
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Heart Failure; Arrhythmias, Cardiac | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Light Chain Cardiac Amyloidosis: Participants with light chain cardiac amyloidosis actively receiving chemotherapy or undergoing autologous bone marrow transplant
  Interventions: Diagnostic Test: Left Atrial Strain Imaging; Diagnostic Test: Electrocardiography

INTERVENTIONS:
Diagnostic Test: Left Atrial Strain Imaging — Two-dimensional, color Doppler, spectral Doppler recordings will be taken from parasternal, apical, subcostal, and modified sections using a Philips Epiq CVx echocardiography device and X5-1 probe. Conventional parameters, additional parameters, and strain analyzes will be performed with speckle tracking echocardiography from these recordings.
  Other Names: TomTec AutoStrain Suite Software; Philips Epiq CVx Echocardiography System; Philips X5-1 3D Echocardiography Probe
Diagnostic Test: Electrocardiography — Electrocardiography will be taken at baseline and the follow-up periods
  Other Names: Mindray BeneHeart R12 ECG system

SUMMARY:
The purpose of this study to assess the longitudinal changes in left atrial strain and supraventricular arrhythmia burden after chemotherapeutic strategies in cardiac light chain amyloidosis.

DETAILED DESCRIPTION:
Light chain (AL) amyloidosis is a disease characterized by localized or systemic accumulation of amyloid fibrils in tissues caused by abnormal folding of light chain immunoglobulins and affecting organ functions. Due to the accumulation of abnormal folding immunoglobulins in the cardiac conduction system, arrhythmia susceptibility has been reported to increase significantly. Atrioventricular blocks and supraventricular arrhythmia are mainly detected among the most common arrhythmia. While these developing supraventricular arrhythmias and atrioventricular blocks in non-amyloidosis diseases result in increased mortality and morbidity, there is insufficient data on cardiac AL amyloidosis treated with chemotherapy. For this reason, this study was planned, and the purpose of this study is to assess the longitudinal changes in left atrial strain and supraventricular arrhythmia burden after chemotherapeutic strategies in cardiac light chain amyloidosis.

After being informed about the study, it is planned to recruit and follow up AL-Amyloidosis patients with cardiac involvement who are currently receiving/planned chemotherapy followed by hematology or who are planned for bone marrow transplantation within one year after obtaining written consent from the patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Patients who give the informed consent
* Patients with cardiac primary light chain amyloidosis or due to multiple myeloma who are newly diagnosed, currently receiving chemotherapeutic treatment, or are scheduled for bone marrow transplantation

Exclusion Criteria:

* A history of myocardial infarction, coronary artery disease, percutaneous coronary intervention and revascularization
* < 18 years old
* A history of severe aortic and mitral valve disease
* Patients who do not give the informed consent
* A history of severe hypertension (SBP>180 mmHg or DBP ≥110 mmHg or the need to use three or more antihypertensive agents)
* Stable coronary artery patients with ischemia data in stress tests (exertion test, myocardial perfusion scintigraphy)
* Presence of non-amyloidosis, systemic, inflammatory or autoimmune disease
* Patients whose cardiac imaging is not interpretable
* Patients whose ECG is not interpretable

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18-90 years with cardiac primary light chain amyloidosis or due to multiple myeloma who are newly diagnosed, currently receiving chemotherapeutic treatment, or are scheduled for bone marrow transplantation will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
The prognostic significance of longitudinal changes in left atrial strain and supraventricular arrhythmia burden after chemotherapy in cardiac light chain amyloidosis | Baseline, and 1st, 3rd, 6th, 12th Month follow-up
  In this study, the effects of treatment strategies on left atrial strain imaging and supraventricular arrhythmia burden and its relationship with mortality and morbidity will be investigated in patients with AL-amyloidosis, who are still under treatment, and newly diagnosed with AL-amyloidosis.

SECONDARY OUTCOMES:
Evaluation of the effects of treatment strategies on arrhythmia burden | Baseline, and 1st, 3rd, 6th, 12th Month follow-up
  By obtaining the serial ECG records, arrhythmia burden will be recorded/

CONTACTS AND LOCATIONS:
Overall Officials: Burçak Kılıçkıran Avcı, Assoc Prof., Study Chair — Istanbul University - Cerrahpasa; Deniz Mutlu, MD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Witteles RM, Liedtke M. AL Amyloidosis for the Cardiologist and Oncologist: Epidemiology, Diagnosis, and Management. JACC CardioOncol. 2019 Sep 24;1(1):117-130. doi: 10.1016/j.jaccao.2019.08.002. eCollection 2019 Sep. PMID 34396169
- [Result] Badano LP, Kolias TJ, Muraru D, Abraham TP, Aurigemma G, Edvardsen T, D'Hooge J, Donal E, Fraser AG, Marwick T, Mertens L, Popescu BA, Sengupta PP, Lancellotti P, Thomas JD, Voigt JU; Industry representatives; Reviewers: This document was reviewed by members of the 2016-2018 EACVI Scientific Documents Committee. Standardization of left atrial, right ventricular, and right atrial deformation imaging using two-dimensional speckle tracking echocardiography: a consensus document of the EACVI/ASE/Industry Task Force to standardize deformation imaging. Eur Heart J Cardiovasc Imaging. 2018 Jun 1;19(6):591-600. doi: 10.1093/ehjci/jey042. PMID 29596561
- [Result] Inoue K, Kawakami H, Akazawa Y, Higashi H, Higaki T, Yamaguchi O. Echocardiographic Assessment of Atrial Function: From Basic Mechanics to Specific Cardiac Diseases. J Cardiovasc Dev Dis. 2022 Feb 27;9(3):68. doi: 10.3390/jcdd9030068. PMID 35323616
- [Result] Hartnett J, Jaber W, Maurer M, Sperry B, Hanna M, Collier P, Patel DR, Wazni OM, Donnellan E. Electrophysiological Manifestations of Cardiac Amyloidosis: JACC: CardioOncology State-of-the-Art Review. JACC CardioOncol. 2021 Oct 19;3(4):506-515. doi: 10.1016/j.jaccao.2021.07.010. eCollection 2021 Oct. PMID 34729522